CLINICAL TRIAL: NCT03534180
Title: A Phase 2 Study of Venetoclax and Romidepsin With Safety Lead-In for Treatment of Relapsed/Refractory Mature T-Cell Lymphomas
Brief Title: Venetoclax and Romidepsin in Treating Patients With Recurrent or Refractory Mature T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18119; NCI-2018-00810 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18119 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2018-05-09; First posted 2018-05-23 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Anaplastic Large Cell Lymphoma; Recurrent Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Refractory Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell | interventions — romidepsin; Depsipeptides; Lactones; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (venetoclax, romidepsin) (Experimental): Patients receive venetoclax PO QD on days 1-28 and romidepsin IV on days 1, 8, and 15. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Romidepsin; Drug: Venetoclax

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Romidepsin — Given IV
  Other Names: Antibiotic FR 901228; Depsipeptide; FK228; FR901228; Istodax; N-[(3S,4E)-3-Hydroxy-7-mercapto-1-oxo-4-heptenyl]-D-valyl-D-cysteinyl-(2Z)-2-amino-2-butenoyl-L-valine, (4->1) Lactone, Cyclic
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies the side effects and best dose of venetoclax and romidepsin to see how well it works in treating patients with mature T-cell lymphoma that has come back (recurrent) or does not respond to treatment (refractory). Venetoclax and romidepsin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of the combination of venetoclax with romidepsin, including the dose ramp-up, in adults with relapsed or refractory mature T-cell lymphoma. (Safety Lead-in) II. To estimate the efficacy as measured by the overall response rate (ORR) of venetoclax in patients with relapsed or refractory mature T-cell lymphoma. (Phase 2)

SECONDARY OBJECTIVES:

I. To evaluate the complete response rate, duration of response, time to response, overall survival and progression free survival associated with venetoclax and romidepsin in relapsed/refractory mature T-cell lymphoma. (Phase 2) II. To further characterize the safety and toxicities of venetoclax and romidepsin combination in relapsed/refractory mature T-cell lymphoma. (Phase 2)

EXPLORATORY OBJECTIVES:

I. To determine BCL2 protein expression in base line treatment tumor samples and correlatieon with response.

II. To determine changes in Bcl-2 gene expression in pre- and post-treatment tumor samples of mature T- cell lymphoma.

OUTLINE: This is a safety lead-in dose-escalation study, followed by a phase II study.

Patients receive venetoclax orally (PO) once daily (QD) on days 1-28 and romidepsin intravenously (IV) on days 1, 8, and 15. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or the legally authorized representative
* Be willing to provide tissue
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Resolution of all acute toxic effects of prior therapy or surgical procedures to Common Terminology Criteria for Adverse Events (CTCAE) grade =< 1 (except alopecia)
* Failed at least 2 prior systemic therapies. For anaplastic large cell lymphoma (ALCL) histologies this must include failure or intolerable side effects of brentuximab vedotin
* Histologically confirmed peripheral T-cell lymphoma (PTCL) as defined by the World Health Organization (WHO) criteria 2016, excluding cutaneous T-cell lymphoma (CTCL); transformed mycosis fungoides is allowed
* Measurable disease defined as:

  * Computed tomography (CT)/magnetic resonance imaging (MRI)/ or positron emission tomography (PET) scan, with at least one nodal site of disease which is 1.5 cm in longest dimension, and/or spleen > 13 cm in vertical length, and/or diffuse enlargement of liver with or without focal nodules (Lugano 2014); extra nodal sites with biopsy proven abnormal lesions are allowed including skin
  * Patients with only bone marrow involvement will be acceptable
* Prior stem cell transplant allowed

  * If allogeneic hematopoietic cell transplantation (HCT) must have recovered from acute toxicity
  * Cannot have active acute or chronic graft versus host disease (GvHD) and must be off immunosuppressive therapies
* Absolute neutrophil count (ANC) >= 1,000/mm^3 (to be performed within 14 days prior to day 1 of protocol therapy)

  * NOTE: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement
  * Exception: Unless documented bone marrow involvement by lymphoma
* Platelets >= 30,000/mm^3 (to be performed within 14 days prior to day 1 of protocol therapy)

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement
  * Exception: Unless documented bone marrow involvement by lymphoma
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (=< 3 x ULN for Gilbert's syndrome or documented hepatic involvement by lymphoma) (to be performed within 14 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) =< 3 x ULN (to be performed within 14 days prior to day 1 of protocol therapy)

  * If hepatic involvement by lymphoma: AST =< 5 x ULN
* Alanine aminotransferase (ALT) =< 3 x ULN (to be performed within 14 days prior to day 1 of protocol therapy)

  * If hepatic involvement by lymphoma: ALT =< 5 x ULN
* Creatinine clearance of >= 50 mL/min per 24 hour urine or the Cockcroft-Gault formula (to be performed within 14 days prior to day 1 of protocol therapy)
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by WOCBP and males of childbearing potential* to use an adequate method of birth control (hormonal contraception is inadequate) or abstain from heterosexual activity for the course of the study through 90 days after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Bcl2 inhibitors
* Any systemic anti-lymphoma therapy, including monoclonal antibody within 28 days or 5 half-lives (whichever is shorter) of initiating protocol therapy
* Radiation and/or surgery (except lymph node or other diagnostic biopsies) within 14 days prior to day 1 of protocol therapy
* Short course systemic corticosteroids for disease control, improvement of performance status or non-cancer indication within 7 days prior to day 1 of protocol therapy; stable ongoing corticosteroid use (i.e. at least 30 days) up to an equivalent dose of 20 mg of prednisone is permissible
* Strong or moderate CYP3A inhibitors within 7 days prior to day 1 of protocol therapy
* Strong or moderate CYP3A inducers within 7 days prior to day 1 of protocol therapy
* P-gp inhibitors within 7 days prior to day 1 of protocol therapy
* Narrow therapeutic index P-gp substrates within 7 days prior to day 1 of protocol therapy
* Any other investigational agent or used an investigational device within 21 days prior to day 1 of protocol therapy
* Prior surgery or gastrointestinal dysfunction that may affect drug absorption (e.g., gastric bypass surgery, gastrectomy)
* Active human immunodeficiency virus (HIV) or hepatitis C virus (HCV) or hepatitis B virus (HBV); subjects who have an undetectable HIV viral load with CD4 > 200 and are on highly active antiretroviral therapy (HAART) medication are allowed; subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment; those who are PCR positive will be excluded; patients who have had hepatitis C but have finished treatment and are PCR negative will be allowed (testing to be done only in patients suspected of having infections or exposures)
* Concurrent malignancy requiring active therapy
* Known central nervous system or meningeal involvement (in the absence of symptoms, investigation into central nervous system involvement is not required)
* Congestive heart failure (CHF) that meets New York Heart Association (NYHA) class II to IV definitions
* Patients with known cardiac abnormalities such as:

  * Congenital long QT syndrome
  * QTc (corrected QT interval on electrocardiogram [ECG]) interval > 480 milliseconds
  * Any cardiac arrhythmia requiring anti-arrhythmic medication
* Patients with a history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest, unless currently addressed with an automatic implantable cardioverter defibrillator (AICD)
* Active infection requiring systemic therapy
* Unable to swallow capsules, has a partial or small bowel obstruction, or has a gastrointestinal condition resulting in a malabsorptive syndrome (e.g. small bowel resection with malabsorption)
* WOCBP: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine M Zain, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - University of Nebraska Medical Center, Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 participants consented to the study. 9 of them became eligible and received the study treatment.
Period: Overall Study
Arm/Group | Treatment (Venetoclax, Romidepsin)
Started | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Venetoclax, Romidepsin)
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 70 [38 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Grade 3 or Above Toxicities
Description: Graded according to Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 5.0. During the first 2 cycles, all grades of toxicity will be collected. After cycle 2, only the highest grade of any toxicity will be collected for each cycle during protocol treatment and for the period of safety follow-up after end of treatment.
Time Frame: Up to 30 days post-treatment, an average of 4 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Venetoclax, Romidepsin)
Number analyzed (Participants) | 9
Participants | 9

2. Secondary Outcome: Overall Survival at 100 Days
Description: Overall survival (OS) was measured from start of the study treatment to death from any cause. OS to be estimated using the product-limit method of Kaplan- Meier with the Greenwood estimator of standard error.
Time Frame: From the start of study treatment up to 100 days
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Treatment (Venetoclax, Romidepsin)
Number analyzed (Participants) | 9
percent probability | 63 [23 to 86]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed up to 30 days post treatment, an average of 4 months. All-Cause Mortality monitored/assessed up to 5 months post treatment.
Arm/Group | Treatment (Venetoclax, Romidepsin)
All-Cause Mortality (participants affected / at risk) | 6/9
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Venetoclax, Romidepsin) (N=9)
Constipation (Gastrointestinal disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Venetoclax, Romidepsin) (N=9)
Anemia (Blood and lymphatic system disorders) | 7 (40)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (3)
Leukocytosis (Blood and lymphatic system disorders) | 2 (4)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
pancytopenia (Blood and lymphatic system disorders) | 1 (1)
pulmonary embolism (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (6)
Blurred vision (Eye disorders) | 1 (1)
Periorbital edema (Eye disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 2 (8)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Fecal incontinence (Gastrointestinal disorders) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (7)
Vomiting (Gastrointestinal disorders) | 3 (4)
Chills (General disorders) | 2 (6)
Edema limbs (General disorders) | 4 (9)
Fatigue (General disorders) | 5 (6)
Fever (General disorders) | 4 (12)
Fluid overload (General disorders) | 1 (1)
Gait disturbance (General disorders) | 2 (2)
Localized edema (General disorders) | 1 (1)
Shortness Of Breath (General disorders) | 1 (1)
Sore tongue (General disorders) | 1 (1)
intermittent lower right quadrant pain (General disorders) | 1 (1)
left shoulder pain (General disorders) | 1 (1)
night sweats (General disorders) | 1 (1)
nose bleeding (General disorders) | 1 (1)
numbness (General disorders) | 1 (1)
stomach discomfort (General disorders) | 1 (1)
tachypnea (General disorders) | 1 (1)
taste appetite disturbed (General disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (5)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Blood bilirubin increased (Investigations) | 3 (9)
Blood lactate dehydrogenase increased (Investigations) | 2 (3)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 2 (12)
Lymphocyte count decreased (Investigations) | 7 (42)
Neutrophil count decreased (Investigations) | 7 (47)
Platelet count decreased (Investigations) | 8 (37)
Weight gain (Investigations) | 1 (2)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 8 (40)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (10)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (7)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (17)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 5 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (7)
Hyponatremia (Metabolism and nutrition disorders) | 7 (20)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (7)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (4)
Lethargy (Nervous system disorders) | 1 (2)
Memory impairment (Nervous system disorders) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Irritability (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (4)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of Breath at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fungal Rash Chest (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (3)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (5)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (61)
Hypotension (Vascular disorders) | 5 (7)
Jaudice (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT03534180/Prot_SAP_000.pdf